CLINICAL TRIAL: NCT04010942
Title: Therapeutic Effect of Vitamin D3 Supplementation to Clomiphene Citrate Resistant Polycystic Ovary Syndrome Women
Brief Title: Vitamin D for Polycystic Ovary Syndrome Clomiphene Resistant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abouelfath Abouelasrar Gad Dawoud, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VitDPcos
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: PCOS; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Metformin; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Active Comparator): Group V : number of 60 women will receive 100000 IU Cholecalciferol Intramuscular every month + 2000 mg Metformin (oral: 2 tablets 1000 per day) for 5 months .
  -after two months from the start:
  Clomiphene citrate 100mg (2 tablets clomid 50mg each per day,from 2nd to 6th day of the cycle ) will be added every month starting from the 3rd month to the 5th month .
  Interventions: Drug: Vit D; Drug: Metformin; Drug: Clomiphene
- Control (Placebo Comparator): Group C: number of 60 patients will receive Metformin 2000mg (oral: 2 tablets1000 mg per day) for months .
  -after two months from the start:
  Clomiphene citrate 100mg (2 tablets clomid 50mg each per day, from 2nd to 6th day of the cycle ) will be added every month starting from the 3rd month to the 5th month .
  Interventions: Drug: Metformin; Drug: Clomiphene

INTERVENTIONS:
Drug: Vit D — Injection
  Other Names: Devarol-S
  Arms: Vitamin D
Drug: Metformin — tablets
  Other Names: Glucophage extended release
Drug: Clomiphene — Tablet
  Other Names: Clomid

SUMMARY:
This study is determining the therapeutic effect of Vitamin D supplements to Pcos clomiphene resistant polycystic ovarian syndrome Women. Half of patients will receive Vitamin D with metformin while other half metformin only. Then both groups start clomiphene for 3 month

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is considered one of the most common endocrine disorders affecting women in their reproductive age. Genetically it is thought to be involving defects in primary cellular control mechanisms resulting in expression of chronic anovulation and androgen excess. Being familial condition , some researches showed it is autosomal dominant while others thought it is complex trait with oligogenic basis.

Diagnosing poly cystic ovary syndrome is based on finding two of three criteria according to Rotterdam consensus 2003 : oligo/anovulation, clinical/ biochemical signs of hyperandrogenism, ultrasound finding of polycystic ovaries. While insulin resistance which affects 50 - 70 % of PCOS patients is considered to be the main reason for hyperandrogenic features, PCOS also leads to various health problems including metabolic disorders (obesity - Diabetes Mellitus - Cardiovascular diseases) in addition to menstrual irregularities and infertility .

In PCOS women there is polymorphism in Vitamin-D receptor (VDR) gene associated with vitamin D level in blood . This gene is isolated from the female reproductive organs . In VDR null mice; uterine hypoplasia, impaired folliculogenesis and infertility is noted . That's why it is thought to be contributing in the genomic regulation of reproduction.

Several studies have investigated the effectiveness of Vitamin D supplementation to PCOS women they found that PCOS women have hypovitaminosis D3 , with increasing evidence that vitamin D affects insulin and glucose metabolism . vitamin D intake in PCOS women may improve hormonal profiles in addition to having anti-inflammatory and anti-oxidant effects . Another study concluded that Vitamin D and calcium supplementation to PCOS women have a positive effect on BMI, follicular maturation, regularity of menses, androgen related symptoms, infertility and insulin resistance . Moreover, Vitamin D has a crucial role in ovulation induction in women with PCOS.

Vitamin D and calcium in combination with metformin have significant effect on menstrual regulation and follicular development.

Insulin sensitizers such as metformin have been extensively investigated in the management of PCOS. Metformin decreases blood glucose levels by enhancing peripheral glucose uptake, decreasing intestinal glucose absorption and suppressing hepatic glucose levels. In anovulatory women with PCOS, metformin decreases insulin levels, luteinizing hormone (LH) production and circulating androgen levels.

Clomiphene citrate is an estrogen agonist and antagonist. It works by competitively binding estrogen receptors in the thalamus and as it remains in place for an extended period of time, it depletes the body's estrogen concentration at the hypothalamic level. As the body perceives low levels of estrogen, gonadotropin-releasing hormone (GnRH) is released which in turn stimulates pituitary release of follicle stimulating hormone ( FSH) which promotes follicular growth and maturation. If pregnancy is not achieved by 3-6 cycles, other treatments should be considered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS as defined by the Rotterdam criteria
* Females age 20-35 years old
* BMI 18-30 kg/m2
* 1ry or secondary infertility
* Clomiphene resistant ( patients didn't - show response: ovulate to dose of 200 mg clomid per day for 3 cycles )
* Willingness to comply with study protocol for 5 months
* Willingness to give written informed consent to participate in the study

Exclusion Criteria:

* Previous metformin intake
* ovarian drilling
* tubal factor as evidenced by hysterosalpingogram or laparoscope
* endometrial pathology ex., polyp
* Myometrial pathology ex., adenomyosis or fibroid
* abnormal semen parameters
* Cushing syndrome
* Hyperprolactinemia
* Adrenal secreting tumor

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Follicle growth and maturation | 11days
  Transvaginal ultrasound will be done every 48 hours at the start from day 10 of the cycle to assess if the follicle reaches 17-19 mm
Change in Follicle growth and maturation at 3rd month | 11 days
  Transvaginal ultrasound will be done every 48 hours at the start from day 10 of the cycle to assess if the follicle reaches 17-19 mm
Change in Follicle growth and maturation at 5th month | 11 days
  Transvaginal ultrasound will be done every 48 hours at the start from day 10 of the cycle to assess if the follicle reaches 17-19 mm

SECONDARY OUTCOMES:
Occurence of Chemical pregnancy occurence | recorded at any time point during the study whenever occurs up to 5 months
  Positive pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Reda MK Ghanem, Lecturer, Study Director — Obstetrics & Gynecology department Faculty of medicine, Ain shams University.; Ahmed MN Hashaad, Professor, Study Director — Obstetrics & Gynecology department - Faculty of medicine, Ain shams University.
Locations (1):
- Ain Shams University Maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 9 months of study completion
Access Criteria: Requestors should sign a data access agreement. And requests will be revised